CLINICAL TRIAL: NCT03724383
Title: Atrial Fibrillation Lifestyle Project
Acronym: ALP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Teddi Orenstein Lyall (Other)
Collaborators: Vancouver Coastal Health (Other Government); Vancouver Coastal Health Research Institute (Other); University of British Columbia (Other)
Responsible Party: Sponsor-Investigator, Teddi Orenstein Lyall, Cardiologist, VCH-Richmond and Clinical Assistant Professor, Department of Medicine, University of British Columbia, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H18-01441; F18-02253 (Other Grant/Funding Number: Vancouver Coastal Health Research Institute)
Record Dates: First submitted 2018-10-01; First posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: Non-permanent atrial fibrillation; Non-valvular atrial fibrillation; Nutrition; Diet; Exercise; Physical Activity; Sleep Apnea; Cardiovascular Risk; Obesity; Hypertension; Diabetes; Risk Factor Management
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity; Sleep Apnea Syndromes; Obesity; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This is a parallel-group randomized controlled trial. Consecutive patients meeting eligibility criteria that are seen for routine cardiology follow-up will be invited to participate in this study. Patients who accept the possibility of diet counseling and exercise program will be randomized and stratified to 'control arm' versus 'intervention arm.' The final study results will be reported after completion of one-year follow up. We will also carry out a mid-study data analysis at six-months. Forty patients will be randomized to control arm and 40 patients randomized to the intervention arm. Intervention will include Phase 1, a six month program including three months of diet counseling combined with home exercise, followed by three months (starting at week 13) of an in-hospital, Cardiac rehabilitation exercise program. Phase 2 of the intervention will include six months of home-based maintenance exercise and diet (starting at week 25). The entire intervention period will be one year.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators involved in analyzing test results or treating patients are blinded to the participant's study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control arm will receive standard care.
- Intervention (Experimental): Participants in the intervention group will receive risk factor management consultations and take part in 1-hour biweekly diet classes and stress management classes for the first 3 months. This will be followed by 3 months of 1-hour biweekly high intensity interval training exercise classes. At the 6-month time point, participants will be prescribed a home based exercise program and will have the option of participating in weekly group walking sessions. During the final 6 months, participants will use a step/activity tracker to track their steps and heart rate.
  Interventions: Behavioral: Risk Factor Management Consult; Behavioral: Diet Classes; Behavioral: Stress Management Classes; Other: Exercise Classes; Other: Home based exercise program

INTERVENTIONS:
Behavioral: Risk Factor Management Consult — Participants may be referred to an Internist to control risk factor management - this may require monthly visits until risk factor targets have been met.
  Arms: Intervention
Behavioral: Diet Classes — Group nutrition sessions delivered two times per week (1 hr each), over a 3 month period (months 0 to 3 of intervention) delivered by a registered dietitian.
  Arms: Intervention
Behavioral: Stress Management Classes — Group sessions delivered two times per week (1 hr each), over a 3 month period (months 0 to 3 of intervention). Techniques taught will include awareness, coping, and relaxation strategies.
  Arms: Intervention
Other: Exercise Classes — Group sessions delivered two times per week (1 hr each), over 3 month period (months 3-6). Classes will include high intensity interval training, resistance training.
  Arms: Intervention
Other: Home based exercise program — The interval and resistance training program will mirror the supervised exercise.
  Arms: Intervention

SUMMARY:
The objectives of the investigators are to demonstrate a reduction in frequency and symptoms of AF and improvements in cardiovascular risk factors following a lifestyle intervention in patients with paroxysmal AF. Participants will be randomized into control or intervention groups. The intervention will receive step trackers, diet counselling, an exercise program, and risk factor modification consultations. Controls will receive step trackers and care as usual. Testing will occur at baseline, six months, and one year.

DETAILED DESCRIPTION:
Sixty percent of cases of non-valvular AF are associated with other modifiable risk factors, including: obesity, diabetes, hypertension, or sleep apnea. Treating modifiable risk factors has been shown to improve morbidity and mortality in patients with AF. Treatment of AF with antiarrhythmic drugs or catheter ablation has not been shown to improve survival. Recently, small cohort studies combining exercise, diet, and antiarrhythmic medications and/or ablation have shown improvements in cardiovascular risk factors and reduction in AF symptoms and frequency.

The aim of this study is to demonstrate a reduction in frequency and symptoms of AF and improvements in cardiovascular risk factors following a lifestyle intervention in patients with paroxysmal AF. This study uses a reproducible intensive supervised cardiac rehabilitation that includes exercise, diet, and risk factor modification for patients with paroxysmal, non-valvular AF. The investigators expect that a lifestyle intervention will show significant improvement in fitness and weight loss and improvements in AF symptoms and frequency, and cardiovascular risk factors when compared to a control group with paroxysmal AF and similar baseline characteristics who do not receive a diet and exercise program.

ELIGIBILITY:
Inclusion Criteria:

1. paroxysmal, non-permanent, non-valvular AF. Patients with high burden of AF will be admitted into the study ahead of low burden patients.

   1. Low burden paroxysmal AF is defined as: ≥4 episodes of AF over the past 24 months; episodes terminate spontaneously within 7 days or via cardioversion within 48 hours of onset.
   2. High burden paroxysmal AF is defined as: ≥ 4 episodes of AF over the past 6 months, with ≥ 2 episodes > 6 hours in duration; episodes terminate spontaneously within 7 days or via cardioversion within 48 hours of onset.
   3. Early persistent AF is defined as: ≥ 2 episodes of AF over the past 24 months; episodes are successfully terminated via cardioversion within 7 days of onset.
2. BMI equal to or greater than 27 kg/m^2, or central obesity using abdominal circumference with ethnic specific values recommended by Canadian diabetes association.
3. one of hypertension or diabetes

Exclusion Criteria:

1. Permanent AF
2. Estimated survival < 2 years
3. Left ventricular ejection fraction < 40%
4. Weight > 300 lbs, treadmill cannot hold greater weights
5. Inability to walk one city block
6. Severe musculoskeletal or neurological problems making them unable to exercise safely
7. New York Heart Association class 3-4 heart failure
8. Severe aortic valve stenosis
9. Prior mitral valve surgery or severe stenosis or regurgitation
10. Hypertrophic cardiomyopathy
11. Patients with illnesses or medications that already cause atrial fibrillation on their own, such as pericarditis, high doses of prednisone, and hyperthyroidism
12. Any other absolute and relative contraindications to exercise testing
13. Inability to speak and understand English
14. In atrial fibrillation at time of baseline testing
15. Defibrillator present

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Changes in frequency of atrial fibrillation | Baseline to 6 months and 1 year
  The frequency of AF will be measured with 48-hour Holter monitor recording, looking at percent of time in AF.
Changes in severity of atrial fibrillation | Baseline to 6 months and 1 year
  Assessed using the Canadian Cardiovascular Society Severity in Atrial Fibrillation Scale (CCS-SAF), and the Atrial Fibrillation Symptom Severity Scale (AFSS).
  The CCS-SAF categorizes severity of atrial fibrillation from Class 0 to Class 4, with 0 being asymptomatic and 4 being severe.
  On the AFSS, individual symptoms attributable to AF are scored on a five-point Likert scale, such that the total AFSS severity score ranges from 0 to 35, with higher scores indicating increased AFSS.
  These two scales will be used simultaneously to inform the severity of Atrial Fibrillation.
Changes in Quality of Life on SF36 | Baseline to 6 months and 1 year
  The 36-item Short Form Survey Instrument (SF36) measures quality of life. Each question is scored on a Likert scale with varying ranges (0-3, 0-5, etc.). Using a score conversion toolkit, the score for each question is converted to a value out of 100, such that lower scores indicate lower quality of life and higher scores indicate a higher quality of life. Those scores out of 100 can be added to get a score out of 3600, but the quality of life is most often reported as a percent.

SECONDARY OUTCOMES:
Changes in number of medications | Baseline and 1 year
  Total number of all anti-arrhythmic agents, anti-hypertensive agents, diabetes and cholesterol lowering medications will be recorded and compared.
Systolic and Diastolic Blood Pressure | Baseline, 6 months, 1 year
  Measured in mmHg.
  For a normal reading, your blood pressure needs to show a top number (systolic pressure) that's between 90 and less than 120 and a bottom number (diastolic pressure) that's between 60 and less than 80.
Hemoglobin A1C | Baseline, 6 months, 1 year
  The hemoglobin A1c test tells you your average level of blood sugar over the past 2 to 3 months. It's also called HbA1c, glycated hemoglobin test, and glycohemoglobin.
  It is reported in percentages.
Body Mass Index | Baseline, 6 months, 1 year
  Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women. BMI is universally expressed in units of kg/m^2.
Waist Circumference | Baseline, 6 months, 1 year
  Waist circumference is an indicator of health risk associated with excess fat around the waist. A waist circumference of 102 centimetres (40 inches) or more in men, or 88 centimetres (35 inches) or more in women, is associated with health problems such as type 2 diabetes, heart disease and high blood pressure
Relative Fat Mass | Baseline, 6 months, 1 year
  Relative Fat Mass (RFM) is a measure for the estimation of overweight or obesity in humans.
  The ratio or the patient's height and waist measurements in meters is multiplied by 20 before being subtracted from a number (shown in bold below) that adjusts for differences in gender and height:
  RFM for adult males: 64 - (20 x height in meters divided waist circumference in meters) RFM for adult females:76 - (20 x height in metres divided by waist circumference in meters)
Low density lipoprotein | Baseline, 6 months, 1 year
  Low-density lipoprotein (LDL) is one of the body's lipoproteins and an important carrier of cholesterol. LDL is an important marker for the risk of developing heart disease.
  LDL cholesterol levels should be less than 100 mg/dL. Levels of 100 to 129 mg/dL are acceptable for people with no health issues but may be of more concern for those with heart disease or heart disease risk factors. A reading of 130 to 159 mg/dL is borderline high and 160 to 189 mg/dL is high.
Apnea hypopnea index | Baseline, 6 months, 1 year
  The Apnea Hypopnea Index (AHI) is the number of apneas or hypopneas recorded during the study per hour of sleep. It is generally expressed as the number of events per hour. Based on the AHI, the severity of obstructive sleep apnea is classified as follows:
  None/Minimal: AHI < 5 per hour Mild: AHI ≥ 5, but < 15 per hour Moderate: AHI ≥ 15, but < 30 per hour Severe: AHI ≥ 30 per hour
Metabolic equivalents (METs) | Baseline, 6 months, 1 year
  Fitness will be classified using metabolic equivalents (METs).
  One MET is defined as the amount of oxygen consumed while sitting at rest and is equal to 3.5 ml O2 per kg body weight x min. The energy cost of an activity can be determined by dividing the relative oxygen cost of the activity (ml O2/kg/min) x by 3.5. This study will measure metabolic equivalents achieved on exercise stress test.
Left Atrial Volume Index | Baseline,1 year
  The Left Atrial Volume Index (LAVI) is the left atrial volume relative to Body Surface Area (BSA), and is reported in mL/m^2.
  Ranges of LAVI Reference Range 16-28 Mildly Abnormal 29-33 Moderately Abnormal 34-39 Severely Abnormal ≥40
Diastolic Function Grade | Baseline, 1 year
  here are four grades of diastolic dysfunction as described below. Echocardiography is the gold standard to diagnose diastolic dysfunction.
  Grade I (impaired relaxation): This is a normal finding and occurs in nearly 100% of individuals by the age of 60.
  Grade II (pseudonormal): This is pathological and results in elevated left atrial pressures.
  Grade III (reversible restrictive): This results in significantly elevated left atrial pressures.
  Grade IV (fixed restrictive): This indicates a poor prognosis and very elevated left atrial pressures.
Left Atrial Pressure | Baseline, 1 year
  Left atrial pressure (LAP) can be estimated by measuring the systolic blood pressure and the maximum mitral regurgitation velocity by spectral Doppler provided that there is no significant gradient across the aortic valve.
  Left Atrial Pressure is reported in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Teddi Orenstein Lyall, MD, Principal Investigator — University of British Columbia
Locations (7):
- Canada (7):
  - Richmond Hospital Cardiac Rehabilitation, Richmond, British Columbia
  - Richmond Health Services, Richmond, British Columbia
  - Garratt Wellness Centre, Richmond, British Columbia
  - Richmond Cardiology Clinic, Richmond, British Columbia
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Live Well Clinic, Vancouver, British Columbia
  - St. Paul's Healthy Heart Program, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorian P, Cvitkovic SS, Kerr CR, Crystal E, Gillis AM, Guerra PG, Mitchell LB, Roy D, Skanes AC, Wyse DG. A novel, simple scale for assessing the symptom severity of atrial fibrillation at the bedside: the CCS-SAF scale. Can J Cardiol. 2006 Apr;22(5):383-6. doi: 10.1016/s0828-282x(06)70922-9. PMID 16639472
- [Background] Dorian P, Jung W, Newman D, Paquette M, Wood K, Ayers GM, Camm J, Akhtar M, Luderitz B. The impairment of health-related quality of life in patients with intermittent atrial fibrillation: implications for the assessment of investigational therapy. J Am Coll Cardiol. 2000 Oct;36(4):1303-9. doi: 10.1016/s0735-1097(00)00886-x. PMID 11028487
- [Background] Hays, R. D.,&Stewart, A. L. (1992). Construct validity of MOS health measures. In A. L. Stewart&J. E. Ware (eds.), Measuring functioning and well-being: The Medical Outcomes Study approach (pp. 325-342), Durham, NC: Duke University Press.
- [Background] Malmo V, Nes BM, Amundsen BH, Tjonna AE, Stoylen A, Rossvoll O, Wisloff U, Loennechen JP. Aerobic Interval Training Reduces the Burden of Atrial Fibrillation in the Short Term: A Randomized Trial. Circulation. 2016 Feb 2;133(5):466-73. doi: 10.1161/CIRCULATIONAHA.115.018220. Epub 2016 Jan 5. PMID 26733609
- [Background] Chugh SS, Havmoeller R, Narayanan K, Singh D, Rienstra M, Benjamin EJ, Gillum RF, Kim YH, McAnulty JH Jr, Zheng ZJ, Forouzanfar MH, Naghavi M, Mensah GA, Ezzati M, Murray CJ. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation. 2014 Feb 25;129(8):837-47. doi: 10.1161/CIRCULATIONAHA.113.005119. Epub 2013 Dec 17. PMID 24345399
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Guo Y, Tian Y, Wang H, Si Q, Wang Y, Lip GYH. Prevalence, incidence, and lifetime risk of atrial fibrillation in China: new insights into the global burden of atrial fibrillation. Chest. 2015 Jan;147(1):109-119. doi: 10.1378/chest.14-0321. PMID 24921459
- [Background] Lee GA, Stub D, Ling H. Atrial fibrillation in the elderly -- not a benign condition. Int Emerg Nurs. 2012 Oct;20(4):221-7. doi: 10.1016/j.ienj.2012.05.003. Epub 2012 Jul 4. PMID 23084510
- [Background] Wolowacz SE, Samuel M, Brennan VK, Jasso-Mosqueda JG, Van Gelder IC. The cost of illness of atrial fibrillation: a systematic review of the recent literature. Europace. 2011 Oct;13(10):1375-85. doi: 10.1093/europace/eur194. Epub 2011 Jul 14. PMID 21757483
- [Background] Stewart S, Murphy NF, Walker A, McGuire A, McMurray JJ. Cost of an emerging epidemic: an economic analysis of atrial fibrillation in the UK. Heart. 2004 Mar;90(3):286-92. doi: 10.1136/hrt.2002.008748. PMID 14966048
- [Background] Macle L, Cairns J, Leblanc K, Tsang T, Skanes A, Cox JL, Healey JS, Bell A, Pilote L, Andrade JG, Mitchell LB, Atzema C, Gladstone D, Sharma M, Verma S, Connolly S, Dorian P, Parkash R, Talajic M, Nattel S, Verma A; CCS Atrial Fibrillation Guidelines Committee. 2016 Focused Update of the Canadian Cardiovascular Society Guidelines for the Management of Atrial Fibrillation. Can J Cardiol. 2016 Oct;32(10):1170-1185. doi: 10.1016/j.cjca.2016.07.591. Epub 2016 Sep 6. PMID 27609430
- [Background] Huxley RR, Lopez FL, Folsom AR, Agarwal SK, Loehr LR, Soliman EZ, Maclehose R, Konety S, Alonso A. Absolute and attributable risks of atrial fibrillation in relation to optimal and borderline risk factors: the Atherosclerosis Risk in Communities (ARIC) study. Circulation. 2011 Apr 12;123(14):1501-8. doi: 10.1161/CIRCULATIONAHA.110.009035. Epub 2011 Mar 28. PMID 21444879
- [Background] Carlsson AC, Wandell P, Sundquist K, Johansson SE, Sundquist J. Effects of prescribed antihypertensives and other cardiovascular drugs on mortality in patients with atrial fibrillation and hypertension: a cohort study from Sweden. Hypertens Res. 2014 Jun;37(6):553-9. doi: 10.1038/hr.2014.32. Epub 2014 Mar 6. PMID 24599014
- [Background] Eshoo S, Ross DL, Thomas L. Impact of mild hypertension on left atrial size and function. Circ Cardiovasc Imaging. 2009 Mar;2(2):93-9. doi: 10.1161/CIRCIMAGING.108.793190. Epub 2009 Jan 26. PMID 19808574
- [Background] Tsang TS, Barnes ME, Bailey KR, Leibson CL, Montgomery SC, Takemoto Y, Diamond PM, Marra MA, Gersh BJ, Wiebers DO, Petty GW, Seward JB. Left atrial volume: important risk marker of incident atrial fibrillation in 1655 older men and women. Mayo Clin Proc. 2001 May;76(5):467-75. doi: 10.4065/76.5.467. PMID 11357793
- [Background] Tsang TS, Barnes ME, Gersh BJ, Bailey KR, Seward JB. Risks for atrial fibrillation and congestive heart failure in patients >/=65 years of age with abnormal left ventricular diastolic relaxation. Am J Cardiol. 2004 Jan 1;93(1):54-8. doi: 10.1016/j.amjcard.2003.09.012. PMID 14697466
- [Background] Wyse DG, Waldo AL, DiMarco JP, Domanski MJ, Rosenberg Y, Schron EB, Kellen JC, Greene HL, Mickel MC, Dalquist JE, Corley SD; Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) Investigators. A comparison of rate control and rhythm control in patients with atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1825-33. doi: 10.1056/NEJMoa021328. PMID 12466506
- [Background] Neumann T, Wojcik M, Berkowitsch A, Erkapic D, Zaltsberg S, Greiss H, Pajitnev D, Lehinant S, Schmitt J, Hamm CW, Pitschner HF, Kuniss M. Cryoballoon ablation of paroxysmal atrial fibrillation: 5-year outcome after single procedure and predictors of success. Europace. 2013 Aug;15(8):1143-9. doi: 10.1093/europace/eut021. Epub 2013 Feb 17. PMID 23419659
- [Background] Miyazaki S, Taniguchi H, Kusa S, Nakamura H, Hachiya H, Hirao K, Iesaka Y. Five-year follow-up outcome after catheter ablation of persistent atrial fibrillation using a sequential biatrial linear defragmentation approach: What does atrial fibrillation termination during the procedure imply? Heart Rhythm. 2017 Jan;14(1):34-40. doi: 10.1016/j.hrthm.2016.08.041. Epub 2016 Aug 30. PMID 27590435
- [Background] Pathak RK, Elliott A, Middeldorp ME, Meredith M, Mehta AB, Mahajan R, Hendriks JM, Twomey D, Kalman JM, Abhayaratna WP, Lau DH, Sanders P. Impact of CARDIOrespiratory FITness on Arrhythmia Recurrence in Obese Individuals With Atrial Fibrillation: The CARDIO-FIT Study. J Am Coll Cardiol. 2015 Sep 1;66(9):985-96. doi: 10.1016/j.jacc.2015.06.488. Epub 2015 Jun 22. PMID 26113406
- [Background] Hong KL, Glover BM. The impact of lifestyle intervention on atrial fibrillation. Curr Opin Cardiol. 2018 Jan;33(1):14-19. doi: 10.1097/HCO.0000000000000470. PMID 29049041
- [Background] Elliott AD, Maatman B, Emery MS, Sanders P. The role of exercise in atrial fibrillation prevention and promotion: Finding optimal ranges for health. Heart Rhythm. 2017 Nov;14(11):1713-1720. doi: 10.1016/j.hrthm.2017.07.001. Epub 2017 Jul 8. PMID 28694186
- [Background] Jonasson D, Irvine S, Starkey S, Su S, Johal R, Sweeney P, et al. SCREENING FOR OBSTRUCTIVE SLEEP APNEA (OSA) IN ATRIAL FIBRILLATION (AF): WHAT'S THE BEST TEST? Can J Cardiol [Internet]. 2017 Oct 1 [cited 2018 Jan 24];33(10):S195.
- [Background] Froelicher V, Myers J. Exercise and the Heart 5th edition. 5th ed. Pioli SF, editor. Philadelphia: Saunders; 2006.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT03724383/Prot_SAP_000.pdf